CLINICAL TRIAL: NCT00210730
Title: An Open Label Randomized Study To Evaluate The Response Rate Of Epoetin Alfa (PROCRIT�) Versus No/Delayed PROCRIT Treatment In Patients With Cancer And Persistent Chemotherapy-Induced Myelosuppression (Anemia)
Brief Title: The Duration Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped early due to slow enrollment.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004591
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Anemia
Keywords: Anemia; Neoplasm; Hemoglobin Level
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to compare the efficacy of epoetin alfa (PROCRITÂ®) administered subcutaneously (sc) once every week (qw) vs. no epoetin alfa (PROCRITÂ®) treatment in patients with cancer who are anemic.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate hematologic response in patients receiving epoetin alfa (PROCRIT®) therapy for persistent chemotherapy-induced myelosuppression (anemia) after completion of chemotherapy administration as compared to patients who do not receive weekly epoetin alfa (PROCRIT®) immediately after cessation of chemotherapy. Further, the duration of treatment necessary to achieve these endpoints will be studied. A No/Delayed epoetin alfa (PROCRIT®) treatment control (whereby patients in the control group will receive epoetin alfa (PROCRIT®) if their Hb decreases to < 10g/dL during the study) will be used to establish the frequency and magnitude of changes in clinical end points that may occur when epoetin alfa (PROCRIT®) treatment is not continued (or started) for patients with residual myelosuppression after chemotherapy administration has ended. A 2:1 randomization will be used to give every patient a greater chance to receive immediate treatment (66.6% epoetin alfa (PROCRIT®) treatment vs. 33.3% No/Delayed epoetin alfa (PROCRIT®) treatment). The study will be powered to show differences between the two groups in hematologic response.

In this study, the hematologic response is defined as the proportion of patients who are transfusion-free and are able to maintain their mean Hb level at >= 11 g/dL during the study without a Hb drop to <= 10 g/dL and/or transfusion.

The study hypothesis was that immediate epoetin alfa (PROCRIT®) treatment would be more effective in treatment of anemia than No/Delayed epoetin alfa (PROCRIT®) treatment in patients with cancer and persistent chemotherapy-induced anemia. Patients will be randomized 2:1 to receive epoetin alf or no epoetin treatment. The starting dose will be 40,000 Units weekly (QW) or the dose they were on prior to the study (30,000-60,000 Units QW). If the Hb level decreases to <= 10 g/dL, PROCRIT will be initiated at a dose of 40,000 Units QW.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-myeloid malignancy
* Baseline hemoglobin value >= 11 g/dL and <= 12 g/dL unrelated to transfusion
* Female patients with reproductive potential must have a negative serum pregnancy test at screening. Patients must have signed an informed consent

Exclusion Criteria:

* Uncontrolled hypertension
* History (within 6 months) of uncontrolled cardiac arrhythmias, or history of pulmonary emboli, deep vein thrombosis, ischemic stroke, other arterial or venous thrombotic events (excluding superficial thromboses), or known history of chronic coagulation disorder
* Transfusion within 28 days prior to first dose
* Planned myelosuppressive chemotherapy or radiation during study and no prior chemotherapy within 8 weeks or radiation within 4 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-06; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is hematologic response, defined as follows: Transfusion free during study, and the average of post baseline Hb values > 11 g/dL without a post baseline Hb < 10 g/dL.

SECONDARY OUTCOMES:
Proportion of patients transfused, time to first transfusion, proportion of patients with two post baseline Hb values > 12 g/dL, mean final Hb, mean lowest Hb, proportion of patients with Hb < 10, weekly Hb, QOL

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An open label, randomized study to evaluate the response rate of PROCRIT (Epoetin alfa) versus no/delayed PROCRIT treatment in patients with cancer and persistent chemotherapy-induced myelosuppression (anemia). — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=601&filename=CR004591_CSR.pdf